CLINICAL TRIAL: NCT00525057
Title: DVT Prophylaxis in Orthopaedic Oncology Patients - A Safety Study
Brief Title: Dalteparin in Preventing DVT in Participants With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2004-0743; NCI-2018-01848 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2004-0743 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-12

CONDITIONS: Bone Sarcoma; Femur Fracture; Lymphoma; Metastatic Neoplasm; Pathologic Fracture; Plasma Cell Myeloma; Soft Tissue Sarcoma
MeSH Terms: conditions — Bone Neoplasms; Femoral Fractures; Lymphoma; Neoplasm Metastasis; Fractures, Spontaneous; Multiple Myeloma; Sarcoma | interventions — Dalteparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (dalteparin) (Experimental): Participants receive dalteparin SC QD starting 12-24 hours after surgery on post-operative day 1 until hospital discharge, about 7-10 days.
  Interventions: Drug: Dalteparin

INTERVENTIONS:
Drug: Dalteparin — Given SC

SUMMARY:
This trial studies how well dalteparin works in preventing deep vein thrombosis (DVT) (blood clots) in participants with cancer. Dalteparin is a blood thinner that can treat blood clots and may prevent them from forming.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of dalteparin as prophylaxis against deep venous thrombosis (DVT) in orthopedic oncology patients.

II. To determine whether there are significantly increased bleeding complications at the surgical site after major oncologic operations in the lower extremity.

OUTLINE:

Participants receive dalteparin subcutaneously (SC) once daily (QD) starting 12-24 hours after surgery on post-operative day 1 until hospital discharge, about 7-10 days.

ELIGIBILITY:
Inclusion Criteria:

* GROUP A
* Metastatic disease, myeloma, lymphoma.
* Pathologic fracture or impending pathologic fracture of the femur.
* Intramedullary rod, plating, cementation, hip arthroplasty, or knee arthroplasty.
* GROUP B
* Primary sarcoma of bone or soft tissue of the lower extremity.
* T2 tumor (> 5 cm by < 20 cm).
* Radical resection of tumor, which may necessitate major bone or soft tissue reconstruction.

Exclusion Criteria:

* Presence of DVT on pre-operative screening ultrasound study.
* Massive tumor (> 20 cm in greatest dimension).
* Amputation of the affected leg as treatment of tumor.
* Estimated blood loss > 2 liters during surgery.
* Surgical drain output > 500 cc of bloody fluid during first 8 hours.
* International normalized ratio (I.N.R.) > 1.3 pre-operatively or > 1.5 post-operatively.
* Platelet count < 100,000 either pre-operatively or post-operatively.
* Indwelling post-operative epidural catheter for pain control.
* History of underlying bleeding disorder, such as hemophilia.
* History of adverse reaction to heparin such as heparin-induced thrombocytopenia.
* Severe liver or renal insufficiency.
* History of hypertensive or diabetic retinopathy.
* History of gastro-intestinal bleeding within 12 months.
* Treatment with warfarin, clopidogrel, aspirin, nonsteroidal antiinflammatory drugs (NSAIDs), low molecular weight heparin (LMWH) or other anti-coagulants for conditions.
* History of stroke.
* Women of child bearing potential having a positive urine or serum pregnancy test (human chorionic gonadotropin [hCG]) at the time of pre-operative evaluation (within 7 days of surgery).
* Women who are breastfeeding.
* Hemoglobin < 8.0 g/dL.
* Platelet count < 100,000/L.
* Alanine aminotransferase > 100 IU/L.
* Aspartate aminotransferase > 100 IU/L.
* Direct bilirubin > 0.5mg/dL.
* Serum creatinine > 2.0 mg/dL.
* Patients taking COX-2 inhibitors.
* Patients who have fragmented mechanical heart valves.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2006-07-07 (Actual); Primary Completion 2020-06-19 (Actual); Study Completion 2020-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Lin, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: July 2006 - December 2010
Pre-assignment Details: A total of 65 participants enrolled into the trial. 15 participants did not meet entry criteria and were excluded.
Groups:
- Interventional (Dalteparin, Metastatic): Received dalteparin 5000 units daily postop, patients with metastatic disease.
- Interventional (Dalteparin, Sarcoma): Received dalteparin 5000 units daily postop, patients with primary sarcomas.
Period: Overall Study
Arm/Group | Interventional (Dalteparin, Metastatic) | Interventional (Dalteparin, Sarcoma)
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interventional (Dalteparin, Metastatic) | Interventional (Dalteparin, Sarcoma) | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 21 | 41
  >=65 years | 5 | 4 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 14 | 16 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 25 | 25 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 25 | 25 | 50
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
Tumor Location [Count of Participants; unit: Participants]
  Femur/Thigh | 22 | 15 | 37
  Tibia/Calf | 0 | 6 | 6
  Popliteal | 3 | 4 | 7
Tumor Type [Count of Participants; unit: Participants]
  Carcinoma | 25 | 0 | 25
  Sarcoma | 0 | 25 | 25
Surgery [Count of Participants; unit: Participants]
  Wide Excision Only | 0 | 20 | 20
  Segmental Reconstruction | 19 | 5 | 24
  Curettage, Internal Fixation | 6 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Post-operative Wound Complications
Description: Our primary outcome was the incidence of post-surgical complications, to include wound dehiscence, infection, and seroma.
Time Frame: 4 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional (Dalteparin, Metastatic) | Interventional (Dalteparin, Sarcoma)
Number analyzed (Participants) | 25 | 25
Participants
  Seroma | 1 | 4
  Wound Infection | 0 | 3
  Wound Dehiscence | 0 | 1

2. Secondary Outcome: Number of Participants With Occurrence of Venous Thromboembolism
Description: A secondary outcome was the occurrence of venous thrombolembolism in the post-operative period, to include both deep venous thrombosis in the lower extremity as well as pulmonary embolism.
Time Frame: 4 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional (Dalteparin, Metastatic) | Interventional (Dalteparin, Sarcoma)
Number analyzed (Participants) | 25 | 25
Participants
  Deep venous thrombosis | 1 | 0
  Pulmonary embolism | 0 | 0

3. Secondary Outcome: Post-Operative Blood Transfusion
Description: The volume of packed red blood cell transfusion in the post-operative period
Time Frame: 4 weeks after surgery
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Interventional (Dalteparin, Metastatic) | Interventional (Dalteparin, Sarcoma)
Number analyzed (Participants) | 25 | 25
mL | 213 [0 to 685] | 271 [0 to 2059]

ADVERSE EVENTS:
Time Frame: 4 weeks after surgery
Arm/Group | Interventional (Dalteparin, Metastatic) | Interventional (Dalteparin, Sarcoma)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/25
Other Adverse Events (participants affected / at risk) | 1/25 | 4/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interventional (Dalteparin, Metastatic) (N=25) | Interventional (Dalteparin, Sarcoma) (N=25)
Thromboembolic event (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Interventional (Dalteparin, Metastatic) (N=25) | Interventional (Dalteparin, Sarcoma) (N=25)
Seroma (Surgical and medical procedures) | 1 | 4
Wound infection (Surgical and medical procedures) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2009-08-19): https://cdn.clinicaltrials.gov/large-docs/57/NCT00525057/Prot_SAP_000.pdf